CLINICAL TRIAL: NCT04097873
Title: Effectiveness of Ultrasonography Visual Biofeedback for Diaphragm Training in Athletes With Non-specific Lumbo-pelvic Pain
Brief Title: Ultrasonography Biofeedback for Diaphragm Training in Athletes With Non-specific Lumbo-pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ultrasonography-PR65/19-UCM
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Ultrasonography; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragm biofeedback reeducation plus inspiratory training (Experimental)
  Interventions: Other: Diaphragm ultrasonography reeducation plus inspiratory training
- Isolated high-intensity inspiratory muscle training (Active Comparator)
  Interventions: Other: Isolated inspiratory training

INTERVENTIONS:
Other: Diaphragm ultrasonography reeducation plus inspiratory training — Diaphragm biofeedback reeducation plus inspiratory training during 6 weeks
  Arms: Diaphragm biofeedback reeducation plus inspiratory training
Other: Isolated inspiratory training — Isolated high-intensity inspiratory muscle training during 8 weeks
  Arms: Isolated high-intensity inspiratory muscle training

SUMMARY:
Objective: To determine the effectiveness of diaphragm visual biofeedback reeducation by ultrasonography in conjunction with high-intensity inspiratory muscle training versus isolated high-intensity inspiratory muscle training in athletes with lumbo-pelvic pain. Methods: A single blinded randomized clinical trial will be carried out. A total sample of 80 athletes with lumbo-pelvic pain will be recruited and randomized into 2 groups: one group will be treated by isolated high-intensity inspiratory muscle training during 8 weeks, and another group will be treated with diaphragm visual biofeedback reeducation by ultrasonography during 6 weeks in conjunction with high-intensity inspiratory muscle training during 8 weeks. Outcome measurements will be diaphragm muscle thickness evaluated by ultrasonography (main outcome measurement), pain intensity, pressure pain threshold, disability, quality of life and respiratory parameters by spirometry, which will be assessed before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Athletes with non-specific lumbopelvic pain during 6 weeks

Exclusion Criteria:

* Neural disorders
* Systemic disorders
* Cognitive disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Diaphragm muscle thickness | Change from Baseline diaphragm muscle thickness at 8 weeks
  Diaphragm muscle thickness in centimeters evaluated by ultrasonography

SECONDARY OUTCOMES:
Pain intensity | Change from Baseline pain intensity at 8 weeks
  Pain intensity scores evaluated by the Visual Analogue Scale from 0 (No pain) to 100 millimeters (Worst pain)
Pressure pain threshold | Change from Baseline pressure pain threshold at 8 weeks
  Pressure pain threshold in kilograms / squared centimeter evaluated by algometer
Disability | Change from Baseline disability at 8 weeks
  Disability scores evaluated by the self-reported Roland-Morris Disability Questionnaire from 0 (no disability) to 24 points (Maximum disability)
Health-related quality of life scores | Change from Baseline health-related quality of life scores at 8 weeks
  Quality of life scores evaluated by the self-reported Medical Outcomes Study Short-Form 36 questionnaire from 0 (lowest health-related quality of life) to 100 (highest health-related quality of life)
Respiratory parameters percentage | Change from Baseline respiratory parameters percentage at 8 weeks
  Respiratory parameters percentage evaluated by spirometry

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Calvo-Lobo C, Almazan-Polo J, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Palomo-Lopez P, Rodriguez-Sanz D, Lopez-Lopez D. Ultrasonography comparison of diaphragm thickness and excursion between athletes with and without lumbopelvic pain. Phys Ther Sport. 2019 May;37:128-137. doi: 10.1016/j.ptsp.2019.03.015. Epub 2019 Mar 28. PMID 30954705
- [Background] Calvo-Lobo C, Painceira-Villar R, Lopez-Lopez D, Garcia-Paz V, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Palomo-Lopez P. Tarsal Tunnel Mechanosensitivity Is Increased in Patients with Asthma: A Case-Control Study. J Clin Med. 2018 Dec 12;7(12):541. doi: 10.3390/jcm7120541. PMID 30545067
- [Background] Calvo-Lobo C, Diez-Vega I, Martinez-Pascual B, Fernandez-Martinez S, de la Cueva-Reguera M, Garrosa-Martin G, Rodriguez-Sanz D. Tensiomyography, sonoelastography, and mechanosensitivity differences between active, latent, and control low back myofascial trigger points: A cross-sectional study. Medicine (Baltimore). 2017 Mar;96(10):e6287. doi: 10.1097/MD.0000000000006287. PMID 28272251